CLINICAL TRIAL: NCT05312021
Title: Selective PDE9 Inhibition With IMR-687 in Adults With Heart Failure With Preserved Ejection Fraction: a Safety and Efficacy Phase 2 Randomized Clinical Study (SP9In-HFpEF)
Brief Title: Selective PDE9 Inhibition With IMR-687 in Adults With Heart Failure With Preserved Ejection Fraction
Acronym: SP9In-HFpEF
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study Termination
Sponsor: Cardurion Pharmaceuticals, Inc. (Industry)
Collaborators: Imara, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMR687-HFP-201; 2021-006535-25 (EudraCT Number)
Record Dates: First submitted 2022-03-08; First posted 2022-04-05 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: heart failure; HFpEF; preserved ejection fraction; IMR-687; PDE9
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- IMR-687 (Experimental): Participants randomly assigned to this arm will take IMR-687 orally with food BID for 16 weeks. IMR-687 dosing will be 300 mg BID for participants weighing less than 100 kg and 400 mg BID for participants weighing 100 kg or more.
  Interventions: Drug: IMR-687
- Placebo (Placebo Comparator): Participants randomly assigned to this arm will take placebo orally with food BID for 16 weeks.
  Interventions: Other: IMR-687 Placebo

INTERVENTIONS:
Drug: IMR-687 — 150 mg and 200 mg tablets
  Arms: IMR-687
Other: IMR-687 Placebo — Matching placebo to IMR-687
  Arms: Placebo

SUMMARY:
This study is to evaluate whether 16 weeks of treatment with IMR-687 is a safe and effective treatment for patients with Heart Failure with Preserved Ejection Fraction (HFpEF). The primary objective is to evaluate whether IMR-687 reduces NT-proBNP compared to placebo in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ≥45 years
* Weight 60 to 160 kg, inclusive
* LVEF ≥45% by echo within 6 months prior to Screening Visit
* Symptoms of HFpEF requiring treatment with a diuretic(s) for at least 30 days prior to Screening
* NYHA class II to IV at the time of Screening
* LV hypertrophy, by echo within 6 months of screening, defined by either LV mass/BSA >95 g/m² for females and 115 g/m² for males or LV mass/m² for males >44 g/m2.7 for females and 48 g/m2.7 for males
* NT-proBNP criteria either ≥300 pg/mL if in sinus rhythm or ≥700 pg/mL if in atrial fibrillation at screening
* Elevated LV filling pressure criteria are defined as ONE OR MORE of the following:

  1. HF hospitalization within 12 months prior to screening
  2. LA enlargement (LA width (diameter) ≥3.8 cm, LA length ≥5.0 cm, LA area ≥20 cm² , LA volume ≥55 mL, or LA volume index >29 mL/m²) within 6 months of screening for a participant in sinus rhythm
  3. Cardiac catheterization with at least one of the following in the 12 months prior to screening: rest LVEDP or PCWP ≥15 mm Hg, exercise PCWP ≥25 mm Hg, or fluid challenge PCWP ≥18 mm Hg
  4. Echocardiogram criteria of one or more within 6 months of screening for a participant in sinus rhythm: E/e' (mean of lateral and septal) >13, E/e' lateral >12, or E/e' septal >14; or for a participant in atrial fibrillation: E/e' septal >11
* For WOCBP: Two negative pregnancy tests and the use of highly effective contraception up to 3 months following end of study

Exclusion Criteria:

* Any prior echocardiographic imaging measurement of LVEF <40%
* Six-minute walk test (6MWT) distance <100 m or >450 m at Screening Visit
* Kansas City Cardiomyopathy Questionnaire (KCCQ) overall summary score of >80
* Major cardiovascular surgery, or urgent percutaneous coronary intervention (PCI) within the 3 months prior to Screening Visit, or an elective PCI within 30 days prior to Screening Visit
* Any clinical event within 6 months prior to Screening Visit that could have reduced the LVEF (eg, myocardial infarction, coronary artery bypass graft) unless an echocardiographic measurement was performed at least 1 month after the event confirming the LVEF to be ≥45%

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Change in NT-proBNP | Baseline to Week 16
  Calculated as the percent change from Baseline to Week 16 in NT-proBNP

SECONDARY OUTCOMES:
To evaluate the safety and tolerability in IMR-687 versus placebo (TEAEs: Treatment-emergent adverse events | Baseline to Week 16
  An adverse event (AE) is an untoward medical occurrence in a subject who received study drug without regard to the possibility of a causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; and any other medically important serious event as judged by the investigator. AEs are considered treatment-emergent if they have started or worsened after the first application of study drug up to 30 days after end of treatment with study drug.
Change in Baseline to Week 16 in the Kansas City Cardiomyopathy Questionnaire overall summary score | Baseline to Week 16
  The Kansas City Cardiomyopathy Questionnaire is a self-administered questionnaire. It contains 23 items, covering physical function, clinical symptoms, social function, self-efficacy and knowledge, and quality of life, each with different Likert scale wording, including limitations, frequency, bother, change in condition, understanding, levels of enjoyment, and satisfaction. Scores are transformed to a range of 0-100, in which higher scores reflect better health status. A positive change from baseline indicates improvement.
NYHA Classification | Baseline to Week 16
  Change from Baseline to Week 16 in NYHA classification
Change in Baseline to Week 16 in Clinical Composite Score | Baseline to Week 16
  The clinical composite score is defined as follows: Improved = participant improved in KCCQ score questionnaire with no major adverse cardiovascular event. Worsened = participant worsened (markedly or moderately) in KCCQ score or experienced a major adverse cardiovascular event. Unchanged = participant had no worsening in KCCQ score with no major adverse cardiovascular event.
Change From Baseline in Echocardiography (ECHO) Parameters: Left Ventricular End (LVE) Diastolic Diameter, LVE Systolic Diameter, Septal End Diastolic Thickness, Posterior LV Wall End Diastolic Thickness, Relative Wall Thickness, Left Atrial Dimension | Baseline to Week 16
  A limited two-dimensional and Doppler ECHO examination will be done to assess ECHO parameters. A negative change from baseline indicates improvement.
Change From Baseline in Echocardiography Parameters: LVE Diastolic Volume, LVE Systolic Volume, Left Ventricular Stroke Volume, Left Atrial Volume | Baseline to Week 16
  A limited two-dimensional and Doppler ECHO examination will be done to assess ECHO parameters. A negative change from baseline indicates improvement.
Change From Baseline in Echocardiography Parameters: Left Ventricular Ejection Fraction | Baseline to Week 16
  A limited two-dimensional and Doppler ECHO examination will be done to assess ECHO parameters. A negative change from baseline indicates improvement.
Change From Baseline in Echocardiography Parameters: Left Ventricular Mass | Baseline to Week 16
  A limited two-dimensional and Doppler ECHO examination will be done to assess ECHO parameters. A negative change from baseline indicates improvement.
Change From Baseline in Echocardiography Parameters: Left Ventricular Mass Index | Baseline to Week 16
  A limited two-dimensional and Doppler ECHO examination will be done to assess ECHO parameters. A negative change from baseline indicates improvement.
Change From Baseline in Echocardiography Parameters: Left Atrial Volume Index | Baseline to Week 16
  A limited two-dimensional and Doppler ECHO examination will be done to assess ECHO parameters. A negative change from baseline indicates improvement.
Change From Baseline in Echocardiography Parameters: Ewave Velocity, A Wave Velocity, e' at Septal Mitral Annulus, e' at Lateral Mitral Annulus | Baseline to Week 16
  A limited two-dimensional and Doppler ECHO examination will be done to assess ECHO parameters. A negative change from baseline indicates improvement.
Change From Baseline in Echocardiography Parameters: Ratio of E to A Velocity, E/e' Ratio | Baseline to Week 16
  A limited two-dimensional and Doppler ECHO examination will be done to assess ECHO parameters. A ratio < 1 indicates improvement.
Change in Echocardiography Parameters: Isovolumic Relaxation Time | Baseline to Week 16
  A limited two-dimensional and Doppler ECHO examination will be done to assess ECHO parameters. A negative change from baseline indicates improvement.
Change From Baseline in Echocardiography Parameters: Tricuspid Regurgitation Velocity | Baseline to Week 16
  A limited two-dimensional and Doppler ECHO examination will be done to assess ECHO parameters. A negative change from baseline indicates improvement.
Exercise Capacity | Baseline to Week 16
  Change from Baseline to Week 16 in 6MWT
Body Composition and Biomarker Measures | Baseline to Week 16
  Change from Baseline to Week 16 for body composition by waist-to-hip ratio, BMI, and Tissue Inhibitor of Metalloproteinases (TIMP)
  Evaluation of TIMP will be performed by central laboratory assessment. A negative change from baseline indicates improvement.
Body Composition and Biomarker Measures | Baseline to Week 16
  Change from Baseline to Week 16 for Procollagen III N-terminal Peptide (PIIINP)
  Evaluation of PIIINP will be performed by central laboratory assessment. A negative change from baseline indicates improvement.
Body Composition and Biomarker Measures | Baseline to Week 16
  Change from Baseline to Week 16 for Matrix Metalloproteinase-2 (MMP-2)
  Evaluation of serum MMP-2 will be performed by central laboratory assessment. A negative change from baseline indicates improvement.
Body Composition and Biomarker Measures | Baseline to Week 16
  Change from Baseline to Week 16 for C-peptide
  Evaluation of serum C-peptide will be performed by central laboratory assessment. A negative change from baseline indicates improvement.
Body Composition and Biomarker Measures | Baseline to Week 16
  Change from Baseline to Week 16 for Interleukin-6 (IL-6)
  Evaluation of serum IL-6 will be performed by central laboratory assessment. A negative change from baseline indicates improvement.
Change from Baseline to Week 16 for Estimated Glomerular Filtration Rate (eGFR) | Baseline to Week 16
  eGFR will be calculated from the serum creatinine concentration determined by central laboratory assessment. A positive change from baseline indicates improvement.
Change from Baseline to Week 16 for Interferon-gamma (Ifn-gamma) | Baseline to Week 16
  Evaluation of serum Ifn-gamma will be performed by central laboratory. A negative change from baseline indicates improvement.
Change from Baseline to Week 16 in body composition quantification by dual-energy X-ray absorptiometry scan (at selected sites) | Baseline to Week 16
  A dual-energy X-ray absorptiometry scan will be done to assess body composition parameters. A negative change indicates improvement

CONTACTS AND LOCATIONS:
Overall Officials: Steve Luperchio, Study Director — Cardurion Pharmaceuticals

IPD SHARING:
Plan to Share IPD: No